CLINICAL TRIAL: NCT02050438
Title: How Total Knee Prosthesis Dessigns Influence in Quality of Live
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Jordi Villalba Modol, Medical Doctor, Corporacion Parc Tauli
Other Study IDs: COTCSPT1JV
Record Dates: First submitted 2014-01-29; First posted 2014-01-30 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Osteoarthritis Knee; Total Knee Replacement
Keywords: Osteoarthritis Knee; Total Knee Arthroplasty; Quality of Life
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Knee Osteoarthritis patients with prostesis treatment: Patients operated previously of Knee Osteoarthritis with different prostesis designs according the Hospital guide
  Interventions: Procedure: Total Knee Arthroplasty

INTERVENTIONS:
Procedure: Total Knee Arthroplasty
  Other Names: Total Knee Prostesis

SUMMARY:
The purpose of this study is to determine whether different kind of prostesis designs influences in the quality of life of patients

DETAILED DESCRIPTION:
Objectiu Criteris d'inclusió Mesura dels resultats

ELIGIBILITY:
Inclusion Criteria:

* Aged 65-80 years.
* Primary Ostheortritis
* Mechanical Axis 0+/- 7 degrees

Exclusion Criteria:

* Patients with any new important disease after the surgical procedure.
* Important complications related with the surgical procedure, as fractures, infections and vascular lesions.
* Patients not following a rehabilitation program

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients operated Total Knee Arthroplasty 6 months previously the observational study
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 6 months

SECONDARY OUTCOMES:
Functional Results | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Villaba-Modol, MD, Principal Investigator — Corporacio Sanitaria Parc Tauli
Locations (1):
- Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain